CLINICAL TRIAL: NCT04942249
Title: Long COVID in Military Organisations
Acronym: LoCoMo
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Collaborators: Labor Speiz (Unknown); Swiss Armed Forces (Other); Universitatsspital Zurich (Unknown)
Responsible Party: Principal Investigator, Patricia Schlagenhauf, Prof. Dr., University of Zurich
Other Study IDs: 2021-00256
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic: 167 symptomatic Swiss army recruits who tested positive for SARS-CoV-2 in 2020
  Interventions: Other: No intervention
- Asymptomatic: 167 asymptomatic Swiss army recruits who tested positive for SARS-CoV-2 in 2020
  Interventions: Other: No intervention
- No evidence of infection: 167 Swiss army recruits with no evidence of infection (who also were tested for SARS-CoV-2 in 2020)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A prospective, longitudinal cohort study designed to follow-up on 500 Swiss military personnel who tested in 2020 for SARS-CoV-2 (regardless of whether positive or negative, but with a known test result). Participants are invited to undergo an intensive test battery to evaluate if they suffer COVID-19 sequelae. The testing will include evaluation of several body systems (cardio-vascular, pulmonary, neurological, ophthalmological, psychological and general) and male fertility in a voluntary subgroup. Immune markers and SARS-CoV-2 reinfection rates will also be evaluated. The study hypothesis is that SARS-CoV-2 infection causes a multi-system disease with sequelae detectable in a significant proportion of army recruits after infection with SARS-CoV-2.

DETAILED DESCRIPTION:
During the COVID-19 pandemic, many members of the Swiss armed forces (SAF) contracted SARS-CoV-2. Up to one fifth may suffer from long-term sequelae, or so-called "Long COVID". The "LoCoMo" study is a prospective, longitudinal cohort study designed to follow-up on 500 tested recruits who tested either positive or negative while serving in the SAF in early 2020.

The aim of this research project is to evaluate long-term sequelae that may have occurred in members of the armed forces. By following up on those army recruits who tested positive and who were either symptomatic or asymptomatic and comparing them with those who test negative; symptoms and sequelae of the infection and impact on life quality can be tracked. The acquired data will also provide insights into the duration of immunity (or lack thereof) after symptomatic and asymptomatic infection and the kinetics of antibody decline in those who test positive. Furthermore, the study allows to follow-up on those army recruits who have confirmed positive tests for SARS-CoV-2 and to compare them to those who were negative. The data collected with this extensive test battery allows for a follow-up on a wide range of symptoms, estimated rates of re-infection as well as long- term sequelae after infection, including impact on ophthalmological function, on life quality and activities and impact on male fertility.

The results of the study can also be extrapolated to health-care workers and other young adults who constitute the backbone of the workforce. Because the proposed test battery is very broad and comprehensive it may also detect hitherto unknown, long-term sequelae, which might provide insight in the pathophysiology and general understanding of consequences of SARS-CoV-2 infection which is the basis to develop strategies to mitigate the sequelae. This study will provide essential knowledge on the multi-organ impact of COVID-19 in young persons in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Army recruits and personnel who tested for SARS-CoV-2.
* Completion of a consent form.
* Willing to participate and to complete the testing day in Zürich.

Additional inclusion criteria solely for the voluntary spermiogram test:

* Male
* No known abnormality of the reproductive system (e.g. Klinefelter-Syndrome)

Exclusion Criteria:

* Unwilling to provide consent. Unable to attend the testing day in Zurich.
* A narrow-angle glaucoma or sensitivity to a component of the Tropicamide eye drops is not an exclusion criterion, but the eye examination will be performed without pharmacological mydriasis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The project population is Swiss army recruits who were tested for SARS-CoV-2 in 2020 (regardless of whether they tested positive or negative, but with a known test result). The total number of participants is 500 stratified to 167 participants per infection status (symptomatic, asymptomatic or no evidence of infection).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
to longitudinally follow-up on a cohort of 500 military who tested either positive or negative for SARS-CoV-2 in early 2020 for possible sequelae, one year post infection | One year
  The primary endpoint is the occurrence of SARS-CoV-2 infection sequelae in a longitudinally follow-up cohort of a total of 500 military who tested either positive or negative for SARS-CoV-2 in early 2020.

SECONDARY OUTCOMES:
Outcomes from components of the test battery | One year
  The test battery will detect anticipated sequelae in the following categories: general systemic, pulmonary, cardiac, male fertility, psychological, ophthalmological.

CONTACTS AND LOCATIONS:
Locations (1):
- Epidemiology, Biostatistics and Prevention Institute at the University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azim D, Nasim S, Kumar S, Hussain A, Patel S. Neurological Consequences of 2019-nCoV Infection: A Comprehensive Literature Review. Cureus. 2020 Jun 24;12(6):e8790. doi: 10.7759/cureus.8790. PMID 32601577
- [Background] Banerjee D, Viswanath B. Neuropsychiatric manifestations of COVID-19 and possible pathogenic mechanisms: Insights from other coronaviruses. Asian J Psychiatr. 2020 Dec;54:102350. doi: 10.1016/j.ajp.2020.102350. Epub 2020 Aug 12. PMID 33271682
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] Battaglini D, Brunetti I, Anania P, Fiaschi P, Zona G, Ball L, Giacobbe DR, Vena A, Bassetti M, Patroniti N, Schenone A, Pelosi P, Rocco PRM, Robba C. Neurological Manifestations of Severe SARS-CoV-2 Infection: Potential Mechanisms and Implications of Individualized Mechanical Ventilation Settings. Front Neurol. 2020 Aug 12;11:845. doi: 10.3389/fneur.2020.00845. eCollection 2020. PMID 32903391
- [Background] Bielecki M, Zust R, Siegrist D, Meyerhofer D, Crameri GAG, Stanga Z, Stettbacher A, Buehrer TW, Deuel JW. Social Distancing Alters the Clinical Course of COVID-19 in Young Adults: A Comparative Cohort Study. Clin Infect Dis. 2021 Feb 16;72(4):598-603. doi: 10.1093/cid/ciaa889. PMID 32594121
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Chen L, Deng C, Chen X, Zhang X, Chen B, Yu H, Qin Y, Xiao K, Zhang H, Sun X. Ocular manifestations and clinical characteristics of 535 cases of COVID-19 in Wuhan, China: a cross-sectional study. Acta Ophthalmol. 2020 Dec;98(8):e951-e959. doi: 10.1111/aos.14472. Epub 2020 May 18. PMID 32421258
- [Background] Del Rio C, Collins LF, Malani P. Long-term Health Consequences of COVID-19. JAMA. 2020 Nov 3;324(17):1723-1724. doi: 10.1001/jama.2020.19719. No abstract available. PMID 33031513
- [Background] Disser NP, De Micheli AJ, Schonk MM, Konnaris MA, Piacentini AN, Edon DL, Toresdahl BG, Rodeo SA, Casey EK, Mendias CL. Musculoskeletal Consequences of COVID-19. J Bone Joint Surg Am. 2020 Jul 15;102(14):1197-1204. doi: 10.2106/JBJS.20.00847. PMID 32675661
- [Derived] Deuel JW, Lauria E, Lovey T, Zweifel S, Meier MI, Zust R, Gultekin N, Stettbacher A, Schlagenhauf P. Persistence, prevalence, and polymorphism of sequelae after COVID-19 in unvaccinated, young adults of the Swiss Armed Forces: a longitudinal, cohort study (LoCoMo). Lancet Infect Dis. 2022 Dec;22(12):1694-1702. doi: 10.1016/S1473-3099(22)00449-2. Epub 2022 Aug 26. PMID 36030795